CLINICAL TRIAL: NCT03606642
Title: SYNergy Stent® System Implantation With Mandatory Intra-VascularUltra-Sound Guidance to Examine the Safety of Cessation of Dual Anti-Platelet Therapy in High Bleeding Risk Patients at One Month
Brief Title: SYNergy Stent® System Implantation With Mandatory Intra-VascularUltra-Sound Guidance and Dual Anti-Platelet Therapy
Acronym: SYNIVUS-DAPT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The DSMC March 16, 2022 reviewed of Interim Analysis and recommendation due to no glaring outcomes found to date.
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNIVUS-DAPT
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Stent Placement
Keywords: Cardiovascular disease; peripheral vascular disease (PVD); Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Cardiovascular Diseases; Peripheral Vascular Diseases; Ischemia | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Therapeutics; Ticagrelor; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: DAPT or Dual Antiplatelet Therapy is a combination of two medications given after a percutaneous coronary intervention (PCI) with a drug eluting stent. The medications used for DAPT are low dose Aspirin (81mg) and one of three (3) antiplatelet medications: ticagrelor (Brilinta), clopidogrel (Plavix) or prasugrel (Effient). Because the patients are considered to be at a high risk for bleeding due to one or a combination of reasons this study is trying to determine if a shorter use of DAPT in combination with the Synergy® stent and an imaging tool called IVUS used during your PCI procedure is safe and effective to reduce the potential for serious bleeding events and early stent thrombosis. The Synergy® stent was chosen because of its enhanced method of healing and reduced inflammation of the artery after placement. The Synergy stent may be a better choice for patients who are at high risk for bleeding and could benefit from a shortened period of DAPT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PCI with 30 day DAPT Therapy (Experimental): Single group of patients undergoing IVUS stent placement for PCI with 30 day DAPT therapy regimen. DAPT therapy consists of Aspirin (325 mg loading dose [if applicable] and 81 mg for maintenance dose) and P2Y12 Inhibitor (INFO ABOUT THE DRUGS)
  Interventions: Drug: Dual Antiplatelet (DAPT) Therapy; Device: The Synergy® stent

INTERVENTIONS:
Drug: Dual Antiplatelet (DAPT) Therapy — DAPT - one of three (3) antiplatelet medications: ticagrelor (Brilinta), clopidogrel (Plavix) or prasugrel (Effient) with Aspirin.
  Aspirin loading dose (LD) = 325 mg. Aspirin maintenance dose (MD) = 81 mg.
  P2Y12 Inhibitor Loading Dose (investigator preference):
  Clopidogrel 600 mg PO x 1 or 75 mg PO daily x 4; Prasugrel 60 mg PO x 1; Ticagrelor 180 mg PO x 1.
  P2Y12 Inhibitor Maintenance Dose (investigator preference):
  Clopidogrel 75 mg PO daily; Prasugrel 10 mg PO daily; Ticagrelor 90 mg PO BID.
  Other Names: Ticagrelor (Brilinta); Clopidogrel (Plavix); Prasugrel (Effient) with Aspirin
Device: The Synergy® stent — IVUS guided stent

SUMMARY:
The purpose of this study is to see if one month of dual antiplatelet therapy (DAPT) combined with the placement of the Synergy® Stent with IVUS (intravascular ultrasound) is safe for patients who are at high risk of bleeding (HBR).

DETAILED DESCRIPTION:
DAPT or Dual Antiplatelet Therapy is a combination of two medications given after a percutaneous coronary intervention (PCI) with a drug eluting stent. DAPT is used to help make the platelets in your blood slick so they don't clump or stick together. If the platelets stick together and form a blood clot in the stent it is called a stent thrombosis and will cause an immediate heart attack or MI.

The medications used for DAPT are low dose Aspirin (81mg) and one of three (3) antiplatelet medications: ticagrelor (Brilinta), clopidogrel (Plavix) or prasugrel (Effient) . The standard length of time to take DAPT after a stent placement is 6 months to 1 year. Dapt is associated with an increased risk of bleeding. Because you are considered to be at a high risk for bleeding due to one or a combination of reasons this study is trying to determine if a shorter use of DAPT in combination with the Synergy® stent and an imaging tool called IVUS used during your PCI procedure is safe and effective to reduce the potential for serious bleeding events and early stent thrombosis.

The Synergy® stent was chosen because of its enhanced method of healing and reduced inflammation of the artery after placement. Because of this the Synergy stent may be a better choice for patients who are at high risk for bleeding and could benefit from a shortened period of DAPT.

Intravascular ultrasound or IVUS provides a visual image of the inside of the coronary artery. It is used in patients undergoing PCI or stent placement for a few reasons; prior to placing the stent it is used to measure the artery's width to select the proper size diameter of a stent, also the length of the blockage to select the appropriate length of the stent and to visualize the amount of narrowing or blockage. After the stent is placed IVUS is used to make sure the stent itself is fully expanded and sits up against the wall of the artery. This is called apposition. If stents are not fully expanded and sit up against the wall of the artery early reblockage may occur. In short the IVUS aids in the ideal placement of the stent.

By using the combination of the Synergy® Stent with the IVUS the expectation is to safely decrease the length of time you take DAPT from 6-12 months to 1 month. With the benefit of decreasing the risk of bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered at high risk for bleeding, defined as meeting one or more of the following criteria at the time of enrollment:
* Greater than or equal to 75 years of age and, in the opinion of the investigator, the risk of bleeding associated with >1 months of DAPT outweighs the benefit,
* need for chronic or lifelong anticoagulation therapy
* history of major bleeding (severe/life threatening or moderate bleeding based on the GUSTO classification) within 12 months of the index procedure,
* history of stroke (ischemic or hemorrhagic),
* renal insufficiency (creatinine ≥2.0 mg/dl) or failure (dialysis dependent),
* platelet count ≥20,000/μLto ≤100,000/μL (microliters)
* In the opinion of investigator, patient is at significant risk of falling
* Patient abuses drugs or alcohol
* Hemoglobin ≤11.0 u/dl 2. Subject must be 18 years of age 3. Subject must be able to take study required dual antiplatelet therapy (1 month of P2Y12 inhibitor and aspirin, 13 months of antiplatelet monotherapy) 4. Subject is willing to comply with all protocol requirements, including agreement to stop taking P2Y12 inhibitor at the 1-month milestone if eligible per protocol 5. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific procedures are performed

Angiographic Inclusion Criteria:

1. Subject must have had implantation of at least one Synergy Stent and the use of Boston Scientific IVUS for guided stent implantation
2. All implanted stents must be post dilated and must meet the following IVUS success criteria:

   * treated lesions in which the stent cross sectional area exceeds the distal reference cross sectional area
   * if the stent cross sectional area is less than the distal reference cross sectional area additional post-dilatation must be performed, followed by IVUS
   * above IVUS criteria must be met after the 2nd post dilatation NOTE: if the IVUS criteria is not met after the 2 post dilatation the patient is excluded
3. Stent procedure performed by an approved investigator
4. Vessel diameter ≥ 2.25 mm and ≤4.0 mm and lesion length ≤34mm
5. Pre-dilatation is up to the discretion of the investigator

Exclusion Criteria:

1. Subject with an indication for the index procedure of acute ST elevation MI (STEMI)
2. Subject with an indication for the index procedure of Non ST elevation MI (NSTEMI), based on the 3rd Universal MI definition
3. Subject with treatment with another coronary stent, other than SYNERGY Stent during the index procedure
4. Subject with a planned staged procedure >7 days following the index procedure. (Note: Planned staged procedures are allowed if performed within 7 days of the index procedure and only when SYNERGY stents are used for both the index and staged procedure). Discontinuation of DAPT should occur 1 month after the last PCI procedure is completed.
5. A staged procedure cannot in a 3rd epicardial vessel if 2 epicardial vessels were treated during the index procedure
6. Subject has a known allergy to: contrast (that cannot be adequately pre-medicated), the SYNERGY Stent system or protocol-required concomitant medications (e.g., everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors and aspirin)
7. Subject previously treated at any time with intravascular brachytherapy
8. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
9. Subject is participating in an investigational drug or device clinical trial that has not reached its primary endpoint (Note: registry, observational, data collection studies are not exclusionary)
10. Subject intends to participate in an investigational drug or device clinical trial within 12 months following the index procedure (Note: registry, observational, data collection studies are not exclusionary)
11. Subject is judged inappropriate for discontinuation from P2Y12 inhibitor use at 1 month, due to another condition requiring chronic P2Y12 inhibitor use

    * if at the 30 day visit, the patient has had a peri-procedural NSTEMI with an enzyme elevation >5% of the upper 99th percentile of either creatine kinase-myocardial band (CK-MB) or Troponin, the patient should not be taken off DAPT
12. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor within 1 month following index procedure
13. Subject is a woman who is pregnant or nursing
14. Subject with a current medical condition with a life expectancy of less than 12 months
15. Subject with implantation of a drug-eluting stent other than SYNERGY Stent within 11 months prior to index procedure
16. Have been previously consented for this trial and screen failed
17. Any other clinically significant comorbidities, which in the judgement of the investigator, could compromise compliance with the protocol, interfere with interpretation of the study results, or predispose the patient to safety risks.

Angiographic Exclusion Criteria:

1. Target lesion(s) is located within a saphenous vein graft or an arterial graft
2. TIMI (Thrombolysis In Myocardial Infarction) flow 0 (total occlusion)
3. Target lesion(s) is located in the left main
4. Potential Target lesion(s) that involve a complex bifurcation (i.e. bifurcation lesion requiring treatment with more than one stent)
5. Thrombus, or possible thrombus, present in the target vessel (by visual estimate)
6. Patients requiring a treatment of more than two native epicardial vessels
7. More than three lesions in two epicardial vessels unless they can be covered in one stent
8. In-stent restenosis of target lesion
9. Treatment of non-target lesions or lesions not treated with a Synergy stent
10. Subject who did not receive Boston Scientific IVUS guided stent implantation and assessment
11. Any target lesion that has not been post dilated and has not had post dilatation IVUS
12. Patients who do not meet the following IVUS success criteria:

    * target lesion(s) in which the stent cross sectional area is less than the distal reference cross sectional area and additional post-dilatation should be performed, followed by repeat IVUS.

NOTE: if the IVUS criteria is not met after the 2nd post dilatation, the patient is excluded

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizik, MD, Principal Investigator — HonorHealth Research Institute
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Massachusetts General Hospital, Corrigan Minehan Heart Center, Boston, Massachusetts
  - Northwell Hospital Systems, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An Interim Analysis was completed on December 10, 2021 (Attachment 3) after the 50th enrolled subject completed the 60 day follow up visit. The DSMC (16MAR2022) reviewed the Interim Analysis and recommended to end the study at interim analysis due to no glaring outcomes from the study. They did not see a need to continue, simply due to other similar studies have been completed for similar devices and the point that DAPT can safely be discontinued for High Risk Bleeding patients has been shown.
Groups:
- PCI With 30 Day DAPT Therapy: Single group of patients undergoing IVUS stent placement for PCI with 30 day DAPT therapy regimen. DAPT therapy consists of Aspirin (325 mg loading dose [if applicable] and 81 mg for maintenance dose) and P2Y12 Inhibitor (INFO ABOUT THE DRUGS)
  Dual Antiplatelet (DAPT) Therapy: DAPT - one of three (3) antiplatelet medications: ticagrelor (Brilinta), clopidogrel (Plavix) or prasugrel (Effient) with Aspirin.
  Aspirin loading dose (LD) = 325 mg. Aspirin maintenance dose (MD) = 81 mg.
  P2Y12 Inhibitor Loading Dose (investigator preference):
  Clopidogrel 600 mg PO x 1 or 75 mg PO daily x 4; Prasugrel 60 mg PO x 1; Ticagrelor 180 mg PO x 1.
  P2Y12 Inhibitor Maintenance Dose (investigator preference):
  Clopidogrel 75 mg PO daily; Prasugrel 10 mg PO daily; Ticagrelor 90 mg PO BID (twice a day).
  The Synergy® stent: IVUS guided stent
Period: Overall Study
Arm/Group | PCI With 30 Day DAPT Therapy
Started | 50
Completed | 45
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: An Interim Analysis was completed on December 10, 2021 (Attachment 3) after the 50th enrolled subject completed the 60 day follow up visit. The DSMC (16MAR2022) reviewed the Interim Analysis and recommended to end the study at interim analysis due to no glaring outcomes from the study. They did not see a need to continue, simply due to other similar studies have been completed for similar devices and the point that DAPT can safely be discontinued for High Risk Bleeding patients has been shown.
Groups:
- PCI With 30 Day DAPT Therapy: Single group of patients undergoing IVUS stent placement for PCI with 30 day DAPT therapy regimen. DAPT therapy consists of Aspirin (325 mg loading dose [if applicable] and 81 mg for maintenance dose) and P2Y12 Inhibitor (INFO ABOUT THE DRUGS)
  Dual Antiplatelet (DAPT) Therapy: DAPT - one of three (3) antiplatelet medications: ticagrelor (Brilinta), clopidogrel (Plavix) or prasugrel (Effient) with Aspirin.
  Aspirin loading dose (LD) = 325 mg. Aspirin maintenance dose (MD) = 81 mg.
  P2Y12 Inhibitor Loading Dose (investigator preference):
  Clopidogrel 600 mg PO x 1 or 75 mg PO daily x 4; Prasugrel 60 mg PO x 1; Ticagrelor 180 mg PO x 1.
  P2Y12 Inhibitor Maintenance Dose (investigator preference):
  Clopidogrel 75 mg PO daily; Prasugrel 10 mg PO daily; Ticagrelor 90 mg PO BID.
  The Synergy® stent: IVUS guided stent
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Age, Customized [Count of Participants; unit: Participants] — Greater than or equal to 75 years of age
  Participants
    Greater than or equal to 75 years of age | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 5
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiac Death
Description: Rate of cardiac death from 1 to 13 months post-index procedure in the "as treated" (eligible for 30 day DAPT cessation) population.
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 3

2. Primary Outcome: Rate of Myocardial Infarction
Description: Rate of myocardial infarction (SCAI definition) from 1 to 13 months post-index procedure in the overall enrolled "intent-to-treat" patient population
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 0

3. Secondary Outcome: Number of Participants With Definite/Probable Stent Thrombosis (ST) Based on Academic Research Consortium (ARC) Definition
Description: Rate of Academic Research Consortium (ARC) definite/probable stent thrombosis (ST) involving SYNERGY Stent® from 1 to 13 months post-index procedure
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Number of Participants With Major Bleeding
Description: Rate of major bleeding (GUSTO severe/life threatening + moderate)
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 4

5. Secondary Outcome: Number of Participants With Ischemia-driven (ID) Target Vessel Revascularization,
Description: Angina Assessment
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 0

6. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: Angina Assessment
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 0

7. Secondary Outcome: Number of Participants With All-Cause Death
Description: Angina Assessment
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 4

8. Secondary Outcome: Number of Participants With All-Cause MI (Myocardial Infarction)
Description: Angina Assessment
Time Frame: 1 to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI With 30 Day DAPT Therapy
Number analyzed (Participants) | 50
Participants | 1

ADVERSE EVENTS:
Time Frame: up to 1 year 3 months
Description: A total of 44 non- serious adverse effects have been reported across all sites. Incidence has been as expected for non-cardiac chest discomfort. Others have been varied throughout the study.
  A total of 93 Moderates adverse effects have been reported across all sites which include some hospitalizations.
Arm/Group | PCI With 30 Day DAPT Therapy
All-Cause Mortality (participants affected / at risk) | 4/50
Serious Adverse Events (participants affected / at risk) | 31/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI With 30 Day DAPT Therapy (N=50)
Frontal cerebral bleed/hemorrhagic stroke (Blood and lymphatic system disorders) | 1
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Progression of Lymphoma (Blood and lymphatic system disorders) | 1
Hematoma - Pelvis (Blood and lymphatic system disorders) | 1
Chest Pain (Cardiac disorders) | 3
coranary artery disease- OM1 (Cardiac disorders) | 1
Cardiac Death (Cardiac disorders) | 1
Tachy Brady Syndrome (Cardiac disorders) | 1
Acute Congestive Heart Failure (Cardiac disorders) | 2 — Left Ventricular (LV) diastolic dysfunction; Chronic
Atrial Fibrillation (Cardiac disorders) | 2 — with rapid ventricular response
Acute decompensated heart failure (Cardiac disorders) | 1
Atherosclerosis (Cardiac disorders) | 1 — right lower extremity
GI Bleed (Gastrointestinal disorders) | 1
Acute Abdominal Pain (Gastrointestinal disorders) | 1
intractable nausea and vomiting (Gastrointestinal disorders) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 1
Intrahepatic duct dilatation (General disorders) | 1
multisystem organ dysfunction (General disorders) | 1
Atypical Chest Pain (General disorders) | 1
Sepsis (Infections and infestations) | 3
pneumonia (Infections and infestations) | 2
SARS-CoV-2 (Infections and infestations) | 1
Abscess (Infections and infestations) | 1 — Left Foot
Cellulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1 — Right Foot Infection
Urinary Tract Infection w/Hematuria (Infections and infestations) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
hyperglycemia (Infections and infestations) | 1
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1
Leg fracture (Musculoskeletal and connective tissue disorders) | 2 — proximal Rt. femur and Left Humerus
carcinosarcoma of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
dizzines (Nervous system disorders) | 1
Tremors (Nervous system disorders) | 1
Acute Pyelonephritis (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Endometrial Thickening (Reproductive system and breast disorders) | 1
Abnormal Vaginal Bleeding (Reproductive system and breast disorders) | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Surgical and medical procedures) | 1 — with claudication
Systemic Inflammatory Syndrome (Vascular disorders) | 1
Ischemic Foot (Vascular disorders) | 1
Occlusion of graft right leg (Surgical and medical procedures) | 1
Peripheral Vascular Disease (Vascular disorders) | 1 — with claudication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI With 30 Day DAPT Therapy (N=50)
Anemia (Blood and lymphatic system disorders) | 7 — normocytic; chronic; post-operative; worsening
bruising (Blood and lymphatic system disorders) | 3
prolonged bleeding (Blood and lymphatic system disorders) | 3 — abrasion; groin; nose
Blood in stool (Gastrointestinal disorders) | 2
Hematuria (Blood and lymphatic system disorders) | 1
subhyaloid hemorrhage (Eye disorders) | 1
neutropenic fever (Blood and lymphatic system disorders) | 1
pancytopenia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
atrial tachycardia (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 2
Elevated Cardiac enzymes (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 2 — orthostatic
Junctional Rhythm (Cardiac disorders) | 1
Angina (Cardiac disorders) | 1
subconjunctival hemorrhage (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 2
abdominal pain (Gastrointestinal disorders) | 3
gastroenteritis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Atypical Chest Pain (General disorders) | 2
root canal (General disorders) | 1
Ground level fall (General disorders) | 3
Ear Fullness (Ear and labyrinth disorders) | 1
pain/leak from gastrointestinal tube site (Gastrointestinal disorders) | 1
Gallstones (Hepatobiliary disorders) | 1
Allergic Reaction (Immune system disorders) | 1 — Swollen eye
Pneumonia (Infections and infestations) | 1
SARS CoV2 (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Pain in extremities (Musculoskeletal and connective tissue disorders) | 5 — left arm; right leg; left hip; right hip; right shoulder
venous statis (Musculoskeletal and connective tissue disorders) | 1 — chronic
Fatigue (Musculoskeletal and connective tissue disorders) | 2
Strain (Musculoskeletal and connective tissue disorders) | 1 — Right Arm
Pain (Musculoskeletal and connective tissue disorders) | 1 — Right upper buttock
Myalgias (Musculoskeletal and connective tissue disorders) | 1 — Lower Extremities
Acute exacerbation of chronic lower back pain (Musculoskeletal and connective tissue disorders) | 1
Xyphoidalgia (Musculoskeletal and connective tissue disorders) | 1
Facial Trauma (Musculoskeletal and connective tissue disorders) | 2 — Laceration; contusion post ground-level fall
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 — post motor-vehicle accident
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 3 — Severe; post-motor vehicle accident
Seizure (Nervous system disorders) | 2
Altered Mental Status (Nervous system disorders) | 1
Closed-head injury (Nervous system disorders) | 1
ureteral sone (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
endometrial hyperplasia (Reproductive system and breast disorders) | 1
endometrial polyps (Reproductive system and breast disorders) | 1
endocervical polyp (Reproductive system and breast disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1
metabolic acidosis (Respiratory, thoracic and mediastinal disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 3
Pedal Edema (Vascular disorders) | 2
Peripheral artery disease (Vascular disorders) | 1
pseudoaneurysm (Vascular disorders) | 1 — right wrist
Fistula (Vascular disorders) | 1 — right wrist

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03606642/Prot_SAP_000.pdf